CLINICAL TRIAL: NCT05064215
Title: Lymphatic Drainage of the Breast, a Retrospective Assessment of Data
Status: Completed | Type: Observational
Sponsor: Dr. Elisabeth Würinger (Other)
Responsible Party: Sponsor-Investigator, Dr. Elisabeth Würinger, Dr. Elisabeth Würinger, Wilhelminenspital Vienna
Organization: Wilhelminenspital Vienna (Other)
Other Study IDs: EK 21-102-VK
Record Dates: First submitted 2021-08-24; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Lymph Drainage of Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- injection behind NAC: in 7 breasts dye was injected behind the nipple areola complex before breast reduction
  Interventions: Procedure: anatomical examination
- Injection into lateral upper quadrant: in 5 breasts dye was injected into upper lateral glandular tissue before breast reduction
  Interventions: Procedure: anatomical examination
- injection into medial upper quadrant: in 2 breasts dye was injected into upper medial glandular tissue before breast reduction
  Interventions: Procedure: anatomical examination

INTERVENTIONS:
Procedure: anatomical examination — After injection of dye, its distribution along lymphatic clearance paths was investigated

SUMMARY:
retrospective evaluation of patients, in whom blue colour was injected into different sites of the breast before breast reduction, to investigate direction and localisation of lymphatic flow. Investigations were performed at the Wilhelminenspital, Vienna, in the years 1998 to 2009.

ELIGIBILITY:
Inclusion Criteria: Patients, who understood and supported the aim of the study and signed the written consent -

Exclusion Criteria: language barriers, patients, who did not understand and support the aim of the study

-

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients, who were operated on breast reduction
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Lymphatic flow is guided by the ligamentous suspension | The ligamentous suspension (horizontal septum, vertical ligaments merging into superficial fascia) is exposed in the course of breast reduction in the technique, that I described usually within about 40 minutes
  colour gathered along horizontal septum

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Würinger, Principal Investigator — Dr. Elisabeth Würinger
Locations (1):
- Elisabeth Wuringer, Vienna, Österreich, Austria

IPD SHARING:
Plan to Share IPD: No